CLINICAL TRIAL: NCT01108198
Title: Treatment of Phimosis With Topical Steroid Cream -Double-blind, Randomized, Placebo-controlled Study in 98 Boys
Brief Title: Treatment of Phimosis With Topical Steroid Cream -Double-blind, Randomized, Placebo-controlled Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oulu (Other)
Responsible Party: M.D. Johanna Rättyä, Oulu University Hospital, Department of Children and Adolescents
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1212
Record Dates: First submitted 2010-04-20; First posted 2010-04-21 (Estimated); Last update posted 2010-04-21 (Estimated); Status verified 2010-04

CONDITIONS: Phimosis
Keywords: phimosis,; non-retractable foreskin; topical steroids; children
MeSH Terms: conditions — Phimosis | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- mometasone furoate cream (Active Comparator): The study patient consecutive patients who were referred to outpatient clinic of Pediatric surgery for surgical treatment of non-retractable foreskin. The study patients were randomized to have either mometasone cream or placebo
  Interventions: Drug: Mometasone furoate cream; Drug: moisturizing cream
- moisturizer (Placebo Comparator)
  Interventions: Drug: Mometasone furoate cream; Drug: moisturizing cream

INTERVENTIONS:
Drug: Mometasone furoate cream — Study cream was applicated once per day for 4-8 weeks.
  Other Names: Elocon; topical steroid cream
Drug: moisturizing cream — study cream was applicated once per day for 4 to 8 weeks
  Other Names: Novalan

SUMMARY:
During last years topical steroid creams have been suggested to be effective treatment for non-retractable foreskin instead of circumcision.

Aim of this study is to investigate the efficacy, safety and persistence of treatment results of a medium potent steroid cream in a double-blind, randomized, placebo-controlled study.

ELIGIBILITY:
Inclusion Criteria:

* non-retractable foreskin requiring treatment

Exclusion Criteria:

* age under six years old, previous operation or steroid treatment for phimosis

Ages: 6 Years to 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2006-10; Primary Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Retractability of foreskin | 4-16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Oulu University Hospital, Department of Children and Adolescents, Oulu, Finland